CLINICAL TRIAL: NCT04009447
Title: Sleep Quality and Mechanisms of Cardiovascular Risks in Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00102036
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Insomnia
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive the Cognitive Behavioral Therapy for Insomnia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (Other): Cognitive Behavioral Therapy for Insomnia (CBT-I) 6 sessions of Cognitive Behavioral Training for Insomnia (1 hour each).
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — 6-week CBT-I therapy to help improve sleep quality

SUMMARY:
The objective of this study is to elucidate the potential mechanisms responsible for the increased risk of cardiovascular disease among patients with hypertension and comorbid insomnia.

DETAILED DESCRIPTION:
The investigators propose to utilize a behavioral intervention to manipulate sleep quality in 150 adults with hypertension and comorbid insomnia, who will receive a 6-week Cognitive Behavioral therapy for Insomnia (CBT-I) intervention, which has been shown to markedly improve sleep quality and promote consolidated sleep in approximately 60% of those treated. A lowering of nighttime blood pressure is one of several proposed mechanisms to be examined.

ELIGIBILITY:
Inclusion Criteria:

* Systolic BP ≥ 130 mm Hg based upon two standardized BP screening assessments
* A current diagnosis of insomnia disorder as defined in the International Classification of Sleep Disorders (ICSD-3); or undiagnosed, but suspected, insomnia disorder that is confirmed at their screening lab visit

Exclusion Criteria:

* Uncontrolled hypertension (screening office BP > 160/100 mm Hg)
* Antihypertensive medication use
* Cardiovascular medications
* Previously diagnosed moderate or severe obstructive sleep apnea
* Severe obesity defined by BMI>40 kg/m2
* Pacemakers
* Atrial fibrillation
* Acute coronary syndrome or coronary revascularization procedure within 6 months of enrollment
* Congestive heart failure
* Identifiable cause of hypertension (e.g., primary hyperaldosteronism, renal artery stenosis, untreated hyper- or hypothyroidism, chronic kidney disease, Cushing's disease, pheochromocytoma, coarctation of the aorta)
* Severe uncorrected valvular heart disease
* Current pregnancy
* Active diagnosis of psychosis, bipolar disorder
* Diabetes
* Severely impaired hearing or speech
* Participation in another interventional study to address insomnia
* Rotating shift workers
* Prominent suicidal or homicidal ideation (as assessed through a clinical interview)
* Psychiatric Hospitalization within the past 12 months
* Alcohol or drug abuse within 12 months
* Exposure-based PTSD treatment
* Dementia
* Unstable comorbid sleep disorder requiring assessment and/or treatment outside of the study protocol
* Medical or psychiatric conditions judged to be the primary cause of insomnia
* Inability to comply with the assessment procedures or inability to provide informed consent.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure during the nighttime sleep period | Baseline, 6 week, 12 week, 6 months post intervention
  Average nighttime blood pressure (mm Hg) measured by 24 hour ambulatory blood pressure monitoring before and after CBT-I
Change in sleep during the nighttime sleep period | Baseline, 6 week, 12 week, 6 months post intervention
  Sleep efficiency (percent-time asleep during the sleep period) measured by sleep diary and actigraphy before and after CBT-I.
Changes in insomnia severity | Baseline, 6 week, 12 week, 6 months post intervention
  Insomnia measured by the Insomnia Severity Index before and after CBT-I.

SECONDARY OUTCOMES:
Change in awake blood pressure | Baseline, 6 week, 12 week, 6 months post intervention
  Average awake blood pressure (mm Hg) measured by 24 hour ambulatory blood pressure monitoring before and after CBT-I
Change in nighttime blood pressure dipping | Baseline, 6 week, 12 week, 6 months post intervention
  Average percent change in blood pressure (mm Hg) from awake to nighttime measured by 24 hour ambulatory blood pressure monitoring before and after CBT-I
Change in vascular endothelial function | Baseline, 6 week, 12 week, 6 months post intervention
  Percent dilation of the brachial artery to reactive hyperemia measured by flow mediated dilation before and after CBT-I
Change in arterial stiffness | 6 week, 6 months post intervention
  Pulse wave velocity (m/s) of the descending aorta measured using the Complior system before and after CBT-I
Change in lipid profile | Baseline, 6 week, 12 week, 6 months post intervention
  Lipids (Total, HDL, LDL, Cholesterol and Triglycerides) from fasting venous blood draw measured before and after CBT-I
Change in nighttime sympathetic nervous system activity | 6 week, 12 week
  Measured by 24 hour urine collection (awake and sleep period collection separated) assayed for catecholamines (epinephrine, norepinephrine) and creatinine before and after CBT-I
Change in cardiac structure | 6 week, 6 months post intervention
  Cardiac left ventricular mass (g m^-2.7) before and after CBT-I
Change in cardiac function | 6 week, 6 months post intervention
  Cardiac left ventricular strain (%) before and after CBT-I
Change in sleep fragmentation during the nighttime sleep period | Baseline, 6 week, 12 week, 6 months post intervention
  Sleep Fragmentation Index measured by actigraphy before and after CBT-I.
Change in subjective sleep quality | Baseline, 6 week, 12 week, 6 months post intervention
  Subjective Sleep Quality measured by Pittsburgh Sleep Quality Index before and after CBT-I.
Change in Office Blood Pressure | Baseline, 6 week, 12 week, 6 months post intervention
  Average office seated blood pressure taken by automated clinic blood pressure monitor after 5 minutes rest and based on the average of 3 readings taken at one minute intervals (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sherwood, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherwood A, Ulmer C, Wu JQ, Blumenthal JA, Herold E, Smith PJ, Koch GG, Johnson K, Viera A, Edinger J, Hinderliter A. Cognitive behavior therapy for insomnia for untreated hypertension with comorbid insomnia disorder: The SLEEPRIGHT clinical trial. J Clin Hypertens (Greenwich). 2024 Apr;26(4):441-447. doi: 10.1111/jch.14763. Epub 2024 Mar 11. PMID 38468418

DOCUMENTS (1):
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT04009447/ICF_000.pdf